CLINICAL TRIAL: NCT03045926
Title: Assessment of Elemental Impurities Level After Chronic Administration of Diosmectite (SMECTA®) in Subjects With Chronic Diarrhoea
Brief Title: Chronic Administration of Diosmectite (SMECTA®) in Subjects With Chronic Diarrhoea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D-FR-00250-108; 2016-002111-18 (EudraCT Number)
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Chronic Functional Diarrhea of Unknown Origin
MeSH Terms: interventions — Smectite; smecta

STUDY DESIGN:
Intervention Model Description: The study is interventional Phase 1 without individual benefit.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diosmectite (Smecta®) (Experimental): 5 weeks of diosmectite 3g, 3 times daily.
  Interventions: Drug: Diosmectite (Smecta®)

INTERVENTIONS:
Drug: Diosmectite (Smecta®)

SUMMARY:
The main purpose of this study is to assess the concentration of elemental impurities in blood and urine after chronic administration of Smecta® in subjects with chronic functional diarrhoea. For exploratory purposes, the potential effects of diosmectite on bowel microbiote composition will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, between 18 and 60 years old inclusive, BMI between 19 and 32 kg/m2 inclusive (minimum body weight of 50 kg at screening).
* Functional chronic diarrhoea defined as loose or watery stools occurring in at least 75% of stools for the last 3 months (with symptom onset at least 6 months before diagnosis).

Exclusion Criteria:

* No history of suspected organic or drug induced cause to chronic diarrhoea.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- PRA Health Sciences, Groningen, Netherlands
- MAC Clinical Research Limited, Manchester, United Kingdom

REFERENCES:
- [Derived] Da Silva K, Guilly S, Thirion F, Le Chatelier E, Pons N, Roume H, Quinquis B, Ehrlich SD, Bekkat N, Mathiex-Fortunet H, Sokol H, Dore J. Long-term diosmectite use does not alter the gut microbiota in adults with chronic diarrhea. BMC Microbiol. 2022 Feb 12;22(1):54. doi: 10.1186/s12866-022-02464-7. PMID 35151268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 subjects with chronic functional diarrhoea were enrolled into this open label study in 2 study centres in the Netherlands and United Kingdom. The first subject started 24 August 2016 and last subject completed 9 May 2017.
Pre-assignment Details: 73 subjects were screened for inclusion in the study, 38 subjects failed screening, and 35 met all the inclusion and none of the exclusion criteria. All 35 subjects received treatment with study medication.
Groups:
- Smecta® Powder: Subjects received Smecta® (3 grams [g] of diosmectite), ingested three times a day, in the morning, at noon and in the evening, every day from Day 1 to Day 35 before meals in the fasting state.
  Subjects were followed up for up to 3 months after the last dose of Smecta® administered on Day 35, up to Day 125.
Period: Overall Study
Arm/Group | Smecta® Powder
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the Safety population which consisted of all subjects who received at least one dose of study medication.
Groups:
- Smecta® Powder: Subjects received Smecta® (3 g of diosmectite), ingested three times a day, in the morning, at noon and in the evening, every day from Day 1 to Day 35 before meals in the fasting state.
  Subjects were followed up for up to 3 months after the last dose of Smecta® administered on Day 35, up to Day 125.
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Blood Lead Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood lead levels (BLL) were defined as the average between the available screening and pre-dose (Day-1) values. Values below the limit of detection (LOD) or below the lower limit of quantification (LLOQ) were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in BLL during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in BLL during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: The Intention-to-Treat (ITT) population consisted of all subjects who received at least one dose of study medication and who had one pre-dose BLL and at least one post-dose BLL. Subjects with data available at the timepoints analysed are presented.
Measure: Mean (95% Confidence Interval); unit: nanograms per millilitre (ng/mL)
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
nanograms per millilitre (ng/mL)
  2 hours post-dose, First Dose Day 1 | 0.120 [-0.823 to 1.063]
  Pre-dose, Second Dose Day 1 | 0.306 [-0.661 to 1.273]
  3 hours post-dose, Second Dose Day 1 | 0.095 [-0.886 to 1.076]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 34
  Pre-dose, Third Dose Day 1 | 0.359 [-0.576 to 1.294]
  3 hours post-dose, Third Dose Day 1 | 0.308 [-0.507 to 1.123]
  6 hours post-dose, Third Dose Day 1 | -0.096 [-0.915 to 0.724]
  Pre-dose, First Dose Day 2 | 0.836 [-0.163 to 1.835]
  Pre-dose, First Dose Day 8 | 2.539 [1.702 to 3.375]
  Pre-dose, First Dose Day 15 | 4.722 [3.581 to 5.863]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 34
  Pre-dose, First Dose Day 22 | 6.094 [4.731 to 7.457]
  Pre-dose, First Dose Day 29 | 6.900 [5.338 to 8.462]
  2 hours post-dose, First Dose Day 35 | 6.866 [5.294 to 8.437]
  Pre-dose, Second Dose Day 35 | 7.379 [5.823 to 8.935]
  3 hours post-dose, Second Dose Day 35 | 6.865 [5.376 to 8.354]
  Pre-dose, Third Dose Day 35 | 7.328 [5.783 to 8.874]
  3 hours post-dose, Third Dose Day 35 | 8.248 [5.187 to 11.310]
  6 hours post-dose, Third Dose Day 35 | 6.876 [5.208 to 8.545]
  Day 36 morning | 7.632 [6.029 to 9.234]
  Day 65 (follow-up) | 3.907 [2.613 to 5.201]
  Day 95 (follow-up) | 1.197 [-0.543 to 2.936]
  Day 125 (End of Study) | -0.101 [-1.633 to 1.431]

2. Secondary Outcome: Mean Change From Baseline in Blood Aluminium Concentrations During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood aluminium concentrations were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in blood aluminium concentrations during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in blood aluminium concentrations during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: The ITT population consisted of all subjects who received at least one dose of study medication and who had one pre-dose BLL and at least one post-dose BLL. Subjects with data available at the timepoints analysed are presented.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  2 hours post-dose, First Dose Day 1: number analyzed (Participants) | 30
  2 hours post-dose, First Dose Day 1 | -14.958 [-30.930 to 1.014]
  Pre-dose, Second Dose Day 1: number analyzed (Participants) | 30
  Pre-dose, Second Dose Day 1 | -6.225 [-28.370 to 15.920]
  3 hours post-dose, Second Dose Day 1: number analyzed (Participants) | 30
  3 hours post-dose, Second Dose Day 1 | -13.708 [-29.841 to 2.425]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 28
  Pre-dose, Third Dose Day 1 | -1.688 [-32.375 to 29.000]
  3 hours post-dose, Third Dose Day 1: number analyzed (Participants) | 30
  3 hours post-dose, Third Dose Day 1 | -9.392 [-28.419 to 9.636]
  6 hours post-dose, Third Dose Day 1: number analyzed (Participants) | 29
  6 hours post-dose, Third Dose Day 1 | -14.181 [-31.092 to 2.730]
  Pre-dose, First Dose Day 2: number analyzed (Participants) | 29
  Pre-dose, First Dose Day 2 | -14.181 [-31.092 to 2.730]
  Pre-dose, First Dose Day 8: number analyzed (Participants) | 29
  Pre-dose, First Dose Day 8 | -11.733 [-30.416 to 6.951]
  Pre-dose, First Dose Day 15: number analyzed (Participants) | 29
  Pre-dose, First Dose Day 15 | -15.474 [-31.996 to 1.048]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 28
  Pre-dose, First Dose Day 22 | -2.884 [-33.668 to 27.900]
  Pre-dose, First Dose Day 29: number analyzed (Participants) | 30
  Pre-dose, First Dose Day 29 | -13.708 [-30.050 to 2.633]
  2 hours post-dose, First Dose Day 35: number analyzed (Participants) | 30
  2 hours post-dose, First Dose Day 35 | -13.708 [-28.874 to 1.457]
  Pre-dose, Second Dose Day 35: number analyzed (Participants) | 30
  Pre-dose, Second Dose Day 35 | -13.708 [-29.841 to 2.425]
  3 hours post-dose, Second Dose Day 35: number analyzed (Participants) | 30
  3 hours post-dose, Second Dose Day 35 | -14.958 [-30.930 to 1.014]
  Pre-dose, Third Dose Day 35: number analyzed (Participants) | 30
  Pre-dose, Third Dose Day 35 | -13.708 [-30.050 to 2.633]
  3 hours post-dose, Third Dose Day 35: number analyzed (Participants) | 30
  3 hours post-dose, Third Dose Day 35 | -7.142 [-30.474 to 16.191]
  6 hours post-dose, Third Dose Day 35: number analyzed (Participants) | 30
  6 hours post-dose, Third Dose Day 35 | -13.708 [-30.050 to 2.633]
  Day 36 morning: number analyzed (Participants) | 30
  Day 36 morning | -14.958 [-30.930 to 1.014]
  Day 65 (follow-up: number analyzed (Participants) | 30
  Day 65 (follow-up | -13.708 [-30.050 to 2.633]
  Day 95 (follow-up): number analyzed (Participants) | 30
  Day 95 (follow-up) | -13.708 [-30.050 to 2.633]
  Day 125 (End of Study): number analyzed (Participants) | 30
  Day 125 (End of Study) | -13.708 [-30.050 to 2.633]

3. Secondary Outcome: Mean Change From Baseline in Blood Arsenic Concentrations During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood arsenic concentrations were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in blood arsenic concentrations during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in blood arsenic concentrations during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  2 hours post-dose, First Dose Day 1 | -0.029 [-0.285 to 0.227]
  Pre-dose, Second Dose Day 1 | -0.003 [-0.305 to 0.300]
  3 hours post-dose, Second Dose Day 1 | -0.067 [-0.302 to 0.168]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 34
  Pre-dose, Third Dose Day 1 | -0.059 [-0.327 to 0.209]
  3 hours post-dose, Third Dose Day 1 | 0.037 [-0.311 to 0.384]
  6 hours post-dose, Third Dose Day 1 | 0.034 [-0.298 to 0.366]
  Pre-dose, First Dose Day 2 | 0.027 [-0.311 to 0.365]
  Pre-dose, First Dose Day 8 | 0.312 [-0.221 to 0.846]
  Pre-dose, First Dose Day 15 | 0.484 [-0.196 to 1.165]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 34
  Pre-dose, First Dose Day 22 | 0.429 [0.020 to 0.837]
  Pre-dose, First Dose Day 29 | 0.640 [-0.189 to 1.469]
  2 hours post-dose, First Dose Day 35 | 0.461 [-0.221 to 1.143]
  Pre-dose, Second Dose Day 35 | 0.462 [-0.244 to 1.169]
  3 hours post-dose, Second Dose Day 35 | 0.415 [-0.225 to 1.055]
  Pre-dose, Third Dose Day 35 | 0.420 [-0.209 to 1.050]
  3 hours post-dose, Third Dose Day 35 | 0.361 [-0.248 to 0.970]
  6 hours post-dose, Third Dose Day 35 | 0.359 [-0.239 to 0.956]
  Day 36 morning | 0.350 [-0.223 to 0.922]
  Day 65 (follow-up) | 0.507 [-0.322 to 1.336]
  Day 95 (follow-up) | 0.295 [-0.381 to 0.972]
  Day 125 (End of Study) | 0.051 [-0.433 to 0.535]

4. Secondary Outcome: Mean Change From Baseline in Blood Barium Concentrations During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood barium concentrations were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in blood barium concentrations during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in blood barium concentrations during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  2 hours post-dose, First Dose Day 1 | 0.229 [-0.095 to 0.552]
  Pre-dose, Second Dose Day 1 | 1.300 [-1.342 to 3.942]
  3 hours post-dose, Second Dose Day 1 | 4.229 [-4.129 to 12.586]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 34
  Pre-dose, Third Dose Day 1 | 0.341 [-0.353 to 1.035]
  3 hours post-dose, Third Dose Day 1 | 0.000 [NA to NA] — The confidence interval was not evaluable as blood barium concentrations were below LOD in the majority of subjects.
  6 hours post-dose, Third Dose Day 1 | 0.371 [-0.194 to 0.937]
  Pre-dose, First Dose Day 2 | 0.114 [-0.118 to 0.347]
  Pre-dose, First Dose Day 8 | 0.114 [-0.118 to 0.347]
  Pre-dose, First Dose Day 15 | 0.340 [-0.351 to 1.031]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 34
  Pre-dose, First Dose Day 22 | 0.471 [0.014 to 0.927]
  Pre-dose, First Dose Day 29 | 0.114 [-0.118 to 0.347]
  2 hours post-dose, First Dose Day 35 | 1.086 [-0.673 to 2.844]
  Pre-dose, Second Dose Day 35 | 0.000 [NA to NA] — The confidence interval was not evaluable as blood barium concentrations were below LOD in the majority of subjects.
  3 hours post-dose, Second Dose Day 35 | 0.229 [-0.095 to 0.552]
  Pre-dose, Third Dose Day 35 | 0.563 [-0.371 to 1.497]
  3 hours post-dose, Third Dose Day 35 | 0.114 [-0.118 to 0.347]
  6 hours post-dose, Third Dose Day 35 | 0.000 [NA to NA] — The confidence interval was not evaluable as blood barium concentrations were below LOD in the majority of subjects.
  Day 36 morning | 6.609 [-5.746 to 18.963]
  Day 65 (follow-up) | 0.660 [-0.466 to 1.786]
  Day 95 (follow-up) | 2.423 [-0.974 to 5.820]
  Day 125 (End of Study) | 3.023 [-0.334 to 6.380]

5. Secondary Outcome: Mean Change From Baseline in Blood Cadmium Concentrations During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood cadmium concentrations were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in blood cadmium concentrations during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in blood cadmium concentrations during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  2 hours post-dose, First Dose Day 1 | 0.017 [-0.018 to 0.053]
  Pre-dose, Second Dose Day 1 | -0.002 [-0.035 to 0.032]
  3 hours post-dose, Second Dose Day 1 | 0.020 [-0.030 to 0.070]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 34
  Pre-dose, Third Dose Day 1 | -0.029 [-0.079 to 0.022]
  3 hours post-dose, Third Dose Day 1 | 0.006 [-0.044 to 0.056]
  6 hours post-dose, Third Dose Day 1 | -0.003 [-0.052 to 0.047]
  Pre-dose, First Dose Day 2 | 0.015 [-0.041 to 0.071]
  Pre-dose, First Dose Day 8 | -0.004 [-0.046 to 0.039]
  Pre-dose, First Dose Day 15 | 0.025 [-0.031 to 0.081]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 34
  Pre-dose, First Dose Day 22 | -0.006 [-0.064 to 0.053]
  Pre-dose, First Dose Day 29 | 0.033 [-0.028 to 0.095]
  2 hours post-dose, First Dose Day 35 | -0.009 [-0.067 to 0.049]
  Pre-dose, Second Dose Day 35 | -0.023 [-0.087 to 0.040]
  3 hours post-dose, Second Dose Day 35 | -0.020 [-0.082 to 0.043]
  Pre-dose, Third Dose Day 35 | -0.009 [-0.066 to 0.049]
  3 hours post-dose, Third Dose Day 35 | -0.038 [-0.111 to 0.035]
  6 hours post-dose, Third Dose Day 35 | -0.025 [-0.094 to 0.044]
  Day 36 morning | -0.035 [-0.103 to 0.033]
  Day 65 (follow-up) | 0.034 [-0.042 to 0.110]
  Day 95 (follow-up) | -0.073 [-0.164 to 0.018]
  Day 125 (End of Study) | -0.110 [-0.208 to -0.013]

6. Secondary Outcome: Mean Change From Baseline in Blood Cobalt Concentrations During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood cobalt concentrations were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in blood cobalt concentrations during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in blood cobalt concentrations during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  2 hours post-dose, First Dose Day 1 | 0.006 [-0.037 to 0.050]
  Pre-dose, Second Dose Day 1 | 0.006 [-0.016 to 0.029]
  3 hours post-dose, Second Dose Day 1 | -0.019 [-0.063 to 0.024]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 34
  Pre-dose, Third Dose Day 1 | -0.007 [-0.052 to 0.039]
  3 hours post-dose, Third Dose Day 1 | 0.019 [-0.015 to 0.054]
  6 hours post-dose, Third Dose Day 1 | 0.019 [-0.024 to 0.063]
  Pre-dose, First Dose Day 2 | 0.019 [-0.032 to 0.070]
  Pre-dose, First Dose Day 8 | 0.032 [-0.018 to 0.082]
  Pre-dose, First Dose Day 15 | 0.084 [0.021 to 0.146]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 34
  Pre-dose, First Dose Day 22 | 0.046 [-0.011 to 0.104]
  Pre-dose, First Dose Day 29 | 0.045 [-0.011 to 0.101]
  2 hours post-dose, First Dose Day 35 | 0.045 [-0.011 to 0.101]
  Pre-dose, Second Dose Day 35 | 0.045 [-0.011 to 0.101]
  3 hours post-dose, Second Dose Day 35 | 0.032 [-0.018 to 0.082]
  Pre-dose, Third Dose Day 35 | 0.019 [-0.024 to 0.063]
  3 hours post-dose, Third Dose Day 35 | 0.045 [-0.011 to 0.101]
  6 hours post-dose, Third Dose Day 35 | 0.032 [-0.018 to 0.082]
  Day 36 morning | 0.019 [-0.024 to 0.063]
  Day 65 (follow-up) | 0.084 [0.021 to 0.146]
  Day 95 (follow-up) | -0.006 [-0.070 to 0.057]
  Day 125 (End of Study) | 0.006 [-0.029 to 0.041]

7. Secondary Outcome: Mean Change From Baseline in Blood Mercury Concentrations During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood mercury concentrations were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in blood mercury concentrations during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in blood mercury concentrations during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  2 hours post-dose, First Dose Day 1: number analyzed (Participants) | 31
  2 hours post-dose, First Dose Day 1 | -0.017 [-0.064 to 0.031]
  Pre-dose, Second Dose Day 1: number analyzed (Participants) | 31
  Pre-dose, Second Dose Day 1 | -0.005 [-0.046 to 0.036]
  3 hours post-dose, Second Dose Day 1: number analyzed (Participants) | 31
  3 hours post-dose, Second Dose Day 1 | -0.013 [-0.058 to 0.032]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 30
  Pre-dose, Third Dose Day 1 | 0.013 [-0.034 to 0.060]
  3 hours post-dose, Third Dose Day 1: number analyzed (Participants) | 31
  3 hours post-dose, Third Dose Day 1 | 0.012 [-0.035 to 0.058]
  6 hours post-dose, Third Dose Day 1: number analyzed (Participants) | 31
  6 hours post-dose, Third Dose Day 1 | -0.020 [-0.098 to 0.058]
  Pre-dose, First Dose Day 2: number analyzed (Participants) | 31
  Pre-dose, First Dose Day 2 | 0.015 [-0.028 to 0.059]
  Pre-dose, First Dose Day 8: number analyzed (Participants) | 31
  Pre-dose, First Dose Day 8 | 0.098 [0.001 to 0.194]
  Pre-dose, First Dose Day 15: number analyzed (Participants) | 31
  Pre-dose, First Dose Day 15 | 0.155 [-0.014 to 0.325]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 29
  Pre-dose, First Dose Day 22 | 0.019 [-0.079 to 0.118]
  Pre-dose, First Dose Day 29: number analyzed (Participants) | 29
  Pre-dose, First Dose Day 29 | -0.041 [-0.156 to 0.075]
  2 hours post-dose, First Dose Day 35: number analyzed (Participants) | 29
  2 hours post-dose, First Dose Day 35 | -0.076 [-0.234 to 0.081]
  Pre-dose, Second Dose Day 35: number analyzed (Participants) | 28
  Pre-dose, Second Dose Day 35 | -0.008 [-0.143 to 0.128]
  3 hours post-dose, Second Dose Day 35: number analyzed (Participants) | 28
  3 hours post-dose, Second Dose Day 35 | -0.046 [-0.197 to 0.105]
  Pre-dose, Third Dose Day 35: number analyzed (Participants) | 28
  Pre-dose, Third Dose Day 35 | -0.085 [-0.224 to 0.055]
  3 hours post-dose, Third Dose Day 35: number analyzed (Participants) | 28
  3 hours post-dose, Third Dose Day 35 | -0.091 [-0.236 to 0.053]
  6 hours post-dose, Third Dose Day 35: number analyzed (Participants) | 28
  6 hours post-dose, Third Dose Day 35 | -0.113 [-0.262 to 0.036]
  Day 36 morning: number analyzed (Participants) | 28
  Day 36 morning | -0.085 [-0.224 to 0.055]
  Day 65 (follow-up): number analyzed (Participants) | 20
  Day 65 (follow-up) | 0.064 [-0.034 to 0.161]
  Day 95 (follow-up): number analyzed (Participants) | 22
  Day 95 (follow-up) | 0.080 [-0.252 to 0.411]
  Day 125 (End of Study): number analyzed (Participants) | 23
  Day 125 (End of Study) | 0.112 [-0.167 to 0.390]

8. Secondary Outcome: Mean Change From Baseline in Blood Nickel Concentrations During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline blood nickel concentrations were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in blood nickel concentrations during the treatment period is presented for the timepoints: 2 hours after the first dose, and prior to and after the second and third doses on Days 1 and 35, prior to the first dose on Days 2, 8, 15, 22 and 29, and on Day 36 in the morning.
  The absolute mean change from baseline in blood nickel concentrations during the post-treatment follow-up period is presented for the timepoints: Day 65, Day 95, and Day 125 (End of Study).
Time Frame: Screening and pre-dose Day -1 up to Day 125.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  2 hours post-dose, First Dose Day 1 | 0.000 [-0.562 to 0.562]
  Pre-dose, Second Dose Day 1 | -0.257 [-0.569 to 0.055]
  3 hours post-dose, Second Dose Day 1 | 0.000 [-0.419 to 0.419]
  Pre-dose, Third Dose Day 1: number analyzed (Participants) | 34
  Pre-dose, Third Dose Day 1 | 0.132 [-0.563 to 0.828]
  3 hours post-dose, Third Dose Day 1 | 0.129 [-0.288 to 0.545]
  6 hours post-dose, Third Dose Day 1 | 0.129 [-0.546 to 0.803]
  Pre-dose, First Dose Day 2 | 0.714 [-0.387 to 1.816]
  Pre-dose, First Dose Day 8 | -0.257 [-0.872 to 0.358]
  Pre-dose, First Dose Day 15 | -0.257 [-0.872 to 0.358]
  Pre-dose, First Dose Day 22: number analyzed (Participants) | 34
  Pre-dose, First Dose Day 22 | 0.265 [-0.307 to 0.837]
  Pre-dose, First Dose Day 29 | 0.000 [-0.773 to 0.773]
  2 hours post-dose, First Dose Day 35 | 0.129 [-0.687 to 0.944]
  Pre-dose, Second Dose Day 35 | -0.257 [-0.812 to 0.298]
  3 hours post-dose, Second Dose Day 35 | -0.386 [-0.993 to 0.221]
  Pre-dose, Third Dose Day 35 | 0.129 [-0.643 to 0.900]
  3 hours post-dose, Third Dose Day 35 | 0.000 [-0.676 to 0.676]
  6 hours post-dose, Third Dose Day 35 | 0.000 [-0.773 to 0.773]
  Day 36 morning | -0.257 [-0.978 to 0.463]
  Day 65 (follow-up) | -0.514 [-1.472 to 0.443]
  Day 95 (follow-up) | 0.643 [-0.475 to 1.761]
  Day 125 (End of Study) | 1.414 [0.198 to 2.630]

9. Secondary Outcome: Mean Change From Baseline in Urine Lead Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine lead levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine lead levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: The ITT population consisted of all subjects who received at least one dose of study medication and who had one pre-dose BLL and at least one post-dose BLL.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | 0.040 [-0.168 to 0.248]
  Day 65 (follow-up) | -0.027 [-0.232 to 0.177]
  Day 95 (follow-up) | -0.001 [-0.144 to 0.141]

10. Secondary Outcome: Mean Change From Baseline in Urine Aluminium Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine aluminium levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine aluminium levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | 0.700 [-0.723 to 2.123]
  Day 65 (follow-up) | -1.400 [-3.382 to 0.582]
  Day 95 (follow-up) | -3.500 [-7.119 to 0.119]

11. Secondary Outcome: Mean Change From Baseline in Urine Arsenic Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine arsenic levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine arsenic levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | -2.694 [-22.005 to 16.618]
  Day 65 (follow-up) | -3.886 [-24.165 to 16.394]
  Day 95 (follow-up) | -2.467 [-22.357 to 17.423]

12. Secondary Outcome: Mean Change From Baseline in Urine Barium Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine barium levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine barium levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | 1.493 [0.917 to 2.070]
  Day 65 (follow-up) | -0.188 [-0.643 to 0.266]
  Day 95 (follow-up) | -0.166 [-0.588 to 0.256]

13. Secondary Outcome: Mean Change From Baseline in Urine Cadmium Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine cadmium levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine cadmium levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | -0.051 [-0.114 to 0.011]
  Day 65 (follow-up) | -0.026 [-0.090 to 0.039]
  Day 95 (follow-up) | 0.000 [-0.075 to 0.075]

14. Secondary Outcome: Mean Change From Baseline in Urine Cobalt Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine cobalt levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine cobalt levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | 0.045 [-0.067 to 0.156]
  Day 65 (follow-up) | 0.019 [-0.073 to 0.111]
  Day 95 (follow-up) | 0.115 [-0.080 to 0.311]

15. Secondary Outcome: Mean Change From Baseline in Urine Mercury Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine mercury levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine mercury levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | -0.049 [-0.117 to 0.020]
  Day 65 (follow-up) | -0.024 [-0.074 to 0.025]
  Day 95 (follow-up) | -0.049 [-0.117 to 0.020]

16. Secondary Outcome: Mean Change From Baseline in Urine Nickel Levels During the Treatment Period and Post-treatment Follow-up Period
Description: Baseline urine nickel levels were defined as the average between the available screening and pre-dose (Day-1) values. Values below the LOD or below the LLOQ were replaced by LOD/2 or LLOQ/2 values.
  The absolute mean change from baseline in urine nickel levels are presented for Day 35 of the treatment period (Visit 7, Week 5), and Day 65 (Visit 8, Week 9) and Day 95 (Visit 9, Week 13) in the post-treatment follow-up.
Time Frame: Screening and pre-dose Day -1 up to Day 95.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Smecta® Powder
Number analyzed (Participants) | 35
ng/mL
  Day 35 | -0.090 [-0.423 to 0.243]
  Day 65 (follow-up) | 0.080 [-0.195 to 0.356]
  Day 95 (follow-up) | 0.401 [0.034 to 0.768]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from Day 1 up to Day 125 (End of Study).
Description: TEAEs are reported for the Safety population which consisted of all subjects who received at least one dose of study medication.
Arm/Group | Smecta® Powder
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 30/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smecta® Powder (N=35)
Headache (Nervous system disorders) | 13 (21)
Dizziness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (9)
Gastroenteritis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (8)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Flatulence (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Onycholasis (Skin and subcutaneous tissue disorders) | 1 (1)
Blood glucose increased (Investigations) | 2 (2)
Transferrin increased (Investigations) | 2 (2)
Blood iron increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Chemical injury (Injury, poisoning and procedural complications) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The validity of the analytical methods for vanadium determination in human whole blood and urine was not demonstrated. Therefore, no result for vanadium concentration in the clinical samples is reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall have the right and title to all documentation, reports, records, data, specimens or other work product generated in connection with the performance of the study. All materials, documents, and information of every kind and description supplied by the sponsor (with the exception of that which is in the public domain), and any sponsor intellectual property shall be the sole and exclusive property of the the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT03045926/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03045926/SAP_001.pdf